CLINICAL TRIAL: NCT00706836
Title: PharmacofMRI of Anxiolytic Medications (Pregabalin)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Murray B. Stein, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: UCSD IRB 060407 - B; R01MH075792 (NIH)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Anxiety Disorders
Keywords: anxiety; functional magnetic resonance imaging; fMRI; pregabalin; Lyrica
MeSH Terms: conditions — Anxiety Disorders | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pregabalin 50 mg (Active Comparator): Pregabalin oral tablets (50 mg)
  Interventions: Drug: Pregabalin 50mg
- Pregabalin 200 mg (Active Comparator): Pregabalin oral tablets (200 mg)
  Interventions: Drug: Pregabalin 200 MG
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin 50mg — One dose of oral pregabalin (50 mg) to be administered one hour prior to fMRI scan
  Other Names: Lyrica
  Arms: Pregabalin 50 mg
Drug: Pregabalin 200 MG — One dose of oral pregabalin (200 mg) to be administered one hour prior to fMRI scan
  Other Names: Lyrica
  Arms: Pregabalin 200 mg
Drug: placebo — One dose of matched oral placebo to be administered one hour prior to fMRI scan
  Arms: Placebo

SUMMARY:
The purpose of this study is to use functional magnetic resonance imaging (fMRI) in healthy controls to examine the acute effects of certain anxiolytic medications on brain function. In this case, the medication pregabalin will be used. The investigators hypothesize that pregabalin (at doses of 50 mg and 200 mg, versus placebo) will yield a reduction in amygdala and insula activity (in a dose-dependent fashion) during emotion processing using fMRI.

DETAILED DESCRIPTION:
Increased amygdala and insula activity have been implicated in neurobiological models of anxiety. Using fMRI, the anxiolytic medication, lorazepam, has previously been found to decrease activation in these areas during the processing of emotional stimuli. This study aims to replicate those results but by using a different medication, pregabalin. An eventual aim of this study, in combination with future studies, is to evaluate the utility of fMRI as a tool to identify anxiolytic function in both established and novel compounds that may be used to treat anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Male, or female (not pregnant or intending to become pregnant during the study)
* Between the ages of 18-30.
* In good general health.
* No specific contraindications to the drug being administered

Exclusion Criteria:

* Subjects with a history of DSM-IV depressive disorder, psychotic disorder, anxiety disorder
* Subjects who meet criteria for substance abuse or dependence within the last 6 months
* Subjects with an positive urine screen for illicit drugs having clinically significant abnormal laboratory, ECG or physical examination findings not resolved by the baseline visit
* Patients who have taken psychotropic drugs or antidepressants (including monoamine oxidase inhibitors, MAOI's) within the last year
* Subjects who are left-handed.
* Subjects suffering suffers from claustrophobia, or phobia for injections or blood
* Magnetic Resonance Imaging related exclusion criteria: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), subjects who have ever been a metal worker/welder; history of eye surgery/eyes washed out because of metal, aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, subjects who are in the first trimester of pregnancy, subjects with an I.U.D. (birth control device), a shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Result] Aupperle RL, Ravindran L, Tankersley D, Flagan T, Stein NR, Simmons AN, Stein MB, Paulus MP. Pregabalin influences insula and amygdala activation during anticipation of emotional images. Neuropsychopharmacology. 2011 Jun;36(7):1466-77. doi: 10.1038/npp.2011.32. Epub 2011 Mar 23. PMID 21430645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects recruited by posted advertisements.
Pre-assignment Details: Subjects determined to be healthy based on physical examination, mental health examination, and routine bloodwork.
Groups:
- All Study Participants: Pregabalin oral tablets (50 mg) Pregabalin oral tablets (200 mg) Placebo
  All participants received all 3 treatments on different days.
  Sequence not available.
Period: Overall Study
Arm/Group | All Study Participants
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 16 healthy subjects (10 male; mean age=23.2±2.6)
Groups:
- All 3 Treatments (Cross-Over Design): Pregabalin oral tablets (50 mg) Pregabalin oral tables (200 mg) Placebo
  All subjects received all 3 treatments on different days.
  Sequence data not available.
Arm/Group | All 3 Treatments (Cross-Over Design)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Effect of Pregabalin (Two Doses) Versus Placebo
Description: Region of Interest (ROI) analysis of contrast of doses (high and low) of pregabalin vs placebo on brain activity at rest and during emotional stimuli using fMRI and clinical scales.
Time Frame: Week 1, 2, 3 (Cross-over Design)
Population: Cross-over design, complete data available for all participants. Total number of participants in study is 16; all subjects received all 3 arms of treatment in randomized order.
Measure: Mean (Standard Error); unit: % signal change L amygdala + anticipn
Groups:
- Pregabalin Low Dose (Crossover): Pregabalin oral tablets (50 mg)
  pregabalin: One dose of oral pregabalin (50 mg) to be administered one hour prior to fMRI scan
- Pregabalin High Dose (Crossover): Pregabalin oral tablets (200 mg)
  pregabalin: One dose of oral pregabalin (200 mg) to be administered one hour prior to fMRI scan
- Placebo (Crossover): Placebo
  placebo: One dose of matched oral placebo to be administered one hour prior to fMRI scan
Arm/Group | Pregabalin Low Dose (Crossover) | Pregabalin High Dose (Crossover) | Placebo (Crossover)
Number analyzed (Participants) | 16 | 16 | 16
% signal change L amygdala + anticipn | 0.6 (0.2) | -0.1 (0.1) | 0.6 (0.2)

ADVERSE EVENTS:
Time Frame: Acute within 2 hours of administration
Description: Single dose acute adverse events
Arm/Group | Pregabalin Low Dose (Crossover) | Pregabalin High Dose (Crossover) | Placebo (Crossover)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 4/16 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin Low Dose (Crossover) (N=16) | Pregabalin High Dose (Crossover) (N=16) | Placebo (Crossover) (N=16)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) — Dizziness or lightheadedness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No